CLINICAL TRIAL: NCT03921268
Title: A Randomized Open Label, 3-period, 3-treatment, Crossover Study to Assess the Effect of Inhalation Device and Formulation on Pharmacokinetics Following a Single Inhaled Dose of AZD1402 in Healthy Subjects
Brief Title: Study to Assess Effect of Device and Formulation on Pharmacokinetics (PK) of AZD1402
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D2912C00001
Record Dates: First submitted 2019-03-15; First posted 2019-04-19 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Dose A estimated delivered single dose of AZD1402 nebuliser solution administered via a nebuliser.
  Interventions: Drug: AZD1402
- Treatment B (Experimental): Dose B estimated delivered single dose of AZD1402 inhalation powder administered via an inhaler.
  Interventions: Drug: AZD1402
- Treatment C (Experimental): Dose C estimated delivered single dose of AZD1402 inhalation powder administered via an inhaler.
  Interventions: Drug: AZD1402

INTERVENTIONS:
Drug: AZD1402 — AZD1402 (PRS-060) is presented as a solution and dry powder for oral inhalation and belongs to a new class of therapeutics, Anticalin® proteins, which are modified lipocalins. AZD1402 is an inhaled IL-4Rα antagonist, which is being developed as controller therapy for asthma.
  Other Names: PRS-060

SUMMARY:
To evaluate and compare the pharmacokinetics profiles of AZD1402 after oral inhalation as an inhalation powder and a nebuliser solution.

To further assess the safety and tolerability of single doses of AZD1402 in healthy volunteers.

To evaluate the taste characteristics of the test formulations.

DETAILED DESCRIPTION:
This study will be a randomized, open-label, 3-period, 3-treatment, single dose, single-center, crossover study. Eighteen healthy male and female subjects will be randomized in this study to ensure that at least 12 subjects are evaluable. A subject will be considered to be evaluable if the subject completes all 3 Treatment Periods with no important protocol deviations. Subjects will be randomized to 1 of 6 treatment sequences and will receive each of the 3 single dose treatments of AZD1402 listed below.

* Treatment A: Dose A estimated delivered dose of AZD1402 nebuliser solution administered via a nebuliser.
* Treatment B: Dose B estimated delivered dose of AZD1402 inhalation powder administered via an inhaler.
* Treatment C: Dose C estimated delivered dose of AZD1402 inhalation powder administered via an inhaler.

The study will comprise of:

* A Screening Period of up to 28 days before the first administration of AZD1402.
* Three Treatment Periods during which subjects will be resident at the Clinical Unit from the day before dosing with AZD1402 (Day -1) until at least 48 hours after dosing and discharged on Day 3.
* A Follow-up Visit 10 to 12 days after the last administration of AZD1402 in Treatment Period 3.

Each Treatment Period will be separated by a minimum washout period of 5 days between doses.

All subjects will sign an Informed Consent Form before they participate in any specific study related procedures. Subjects will attend a Screening Visit within 28 days before receiving their first dose of AZD1402. If they are eligible, they will return for Treatment Period 1 when they will have baseline assessments and receive 1 of 3 treatments in a randomized order. For each Treatment Period, the subjects will receive a single dose of Investigational Medicinal Product (IMP) in the morning of Day 1 and have further assessments for 48 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and at Day -1 of Treatment Period 1, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria.

   3.1. Postmenopausal defined as amenorrhea for 2 years or more following cessation of all exogenous hormonal treatments and folliclestimulating hormone (FSH) levels in the postmenopausal range at the Screening Visit.

   3.2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy.

   3.3. Bilateral Tubal ligation at least 5 years prior to the Screening Visit with no subsequent pregnancies.
4. Have a body mass index (BMI) between 18 and 35 kg/m2 inclusive and weigh at least 50 kg.
5. Must be able to demonstrate proper inhalation technique using the Aerosol Inhalation Monitor (AIM) device at the Screening Visit.
6. Subjects must be able to perform reliable spirometry testing according to American Thoracic Society (ATS)/ European Respiratory Society (ERS) criteria at the Screening Visit.
7. Provision of signed, written and dated informed consent for optional genetic research. If a subject decline to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. Subjects who have a significant history of recurrent or ongoing 'dry eye syndrome' of any cause that may be chronic or acute, that may affect the interpretation of safety data associated with the potential for anti-drug antibodies targeted to AZD1402 (structurally related to Tlc).
2. History or clinical manifestations of any clinically significant medical disorder that, in the opinion of the Investigator, may put the subject at risk because of participation in the study, influence the results of the study or affect the subject's ability to participate in the study.
3. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
4. Any clinically significant illness, infection, medical/ surgical procedure, or trauma within 4 weeks of Day 1 of Treatment Period 1, or planned inpatient surgery or hospitalization during the study period.
5. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, at the Screening Visit and/or on Day - 1 of Treatment Period 1, as judged by the PI.
6. Any clinically significant abnormal findings in vital signs at the Screening Visit and/or on Day -1 of Treatment Period 1, as judged by the PI.
7. Any clinically significant abnormalities on 12-lead ECG at the Screening Visit., as judged by the PI.
8. History of, or known significant infection including helminth, hepatitis A, B, or C, HIV, TB (i.e., positive result for interferon (INF) gamma release assay (IGRA), QuantiFERON TB-Gold), that may put the subject at risk during participation in the study.
9. Subjects with history of latent or active TB.
10. Subjects with any history of malignancy or neoplastic disease.
11. Subjects with a disease history suggesting abnormal immune function.
12. History of anaphylaxis following any biologic therapy and known history of allergy or reaction to any component of the investigational product formulation.
13. Subjects who are not able to perform correct spirometry tests at the Screening Visit.
14. Subjects with a forced expiratory volume in the first second (FEV1) and forced vital capacity (FVC) < 80% of the predicted (calculated) values and FEV1/FVC ratio < 0.7 in pulmonary function test (spirometry) at the Screening Visit.
15. Males who are sexually active with a female partner of childbearing potential and who have not had a vasectomy and who do not agree to comply with highly effective methods of contraception from Day 1 of Treatment Period 1 until 90 days after the last dose of IMP.
16. Participation in any clinical study for new chemical entity within the previous 16 weeks or a marketed drug clinical study within the previous 12 weeks or within 5 half-lives whichever is the longer before the first dose of study drug. Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
17. Known or suspected history of drug abuse in the last 5 years
18. Known or suspected history of alcohol abuse or excessive intake of alcohol in the last 2 years
19. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to the Screening Visit.
20. Positive screen for drugs of abuse, alcohol or cotinine at the Screening Visit or on each admission to Clinical Unit.
21. Plasma donation within 1 month of screening or any blood donation/loss more than 450 mL during the 3 months prior to the Screening Visit.
22. Subjects who have received live or attenuated vaccine in the 4 weeks prior to Day 1 of Treatment Period 1.
23. Use of any prescribed or non-prescribed medication including antacids, herbal remedies, megadose vitamins and minerals during the 2 weeks prior to the first administration of IMP or within 5 half-lives whichever is the longer before the first dose of study drug.
24. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives
25. Subjects who have previously received AZD1402.
26. Judgment by the PI that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
27. Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function).
28. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order. In addition, the following is considered a criterion for the exclusion from the optional genetic component of the study
29. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection or previous bone marrow transplant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Area under serum concentration-time curve from zero to infinity [AUC] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the pharmacokinetics (PK) profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Area under the serum concentration-time curve from zero to infinity divided by dose [AUC/D] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Area under the serum concentration-curve from time zero to time of last quantifiable concentration [AUClast] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration divided by dose [AUClast/D] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Maximum observed serum concentration [Cmax] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Observed maximum serum concentration divided by the dose administered [Cmax/D] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Time to reach maximum observed serum concentration [tmax] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Terminal elimination rate constant [λz] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve [t½z] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity [MRT] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Apparent total body clearance of drug from serum after extravascular administration [CL/F] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.
Apparent volume of distribution during the terminal phase after extravascular administration [Vz/F] | Pharmacokinetic Blood Sampling : Day 1: Pre-dose and 5, 20, 40minutes, and 1, 2, 3, 4, 6, 8, 12, 15 and 18 hours post-dose Day 2: 24 and 36 hours postdose. Day 3: 48 hours post-dose
  To evaluate and compare the PK profiles of AZD1402 after oral inhalation as an inhalation powder administered using the Plastiape Monodose inhaler and a nebuliser solution administered using the InnoSpire Go nebuliser.

SECONDARY OUTCOMES:
Number of patients with adverse events | Spontaneous plus Day 1: Pre-dose and 3 and 12 hours post-dose, Day 2: 24 hours post-dose, Day 3: 48 hours post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal findings in vital signs | Day 1: Pre-dose and 10 minutes post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
  Vital signs including BP and Pulse
Number of patients with abnormal electrocardiograms | Day 1: pre-dose and 5 hours post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal physical examination | Day 3: 48 hours post-dose (brief)
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal findings in spirometry | Day 1: pre-dose and 0.5 and 1 hour post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal findings in hematology | Day 3: 48 hours post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal findings in clinical chemistry | Day 3: 48 hours post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Number of patients with abnormal findings in urinalysis | Day 3: 48 hours post-dose
  To further assess the safety and tolerability of single inhaled doses of AZD1402 in healthy volunteers.
Standardized taste questionnaires | Day 1 to Day 3.
  To evaluate the taste characteristics of the test formulations. This will be done immediately after dosing (within 5 minutes). The taste score will be based on 6 attributes: Sweet, Salty, Sour, Bitter, Metallic and Hot/Spicy. Each attribute is with a scale of 0 to 10, where 0= "extremely low/not at all" and 10= "extremely high". If the test formulation is having a smell, another 0 to 10 scale will be there for smell with 0= "extremely bad" and 10= "extremely nice". There will be one score scale with 0="I dislike it extremely much" and 10="I like it extremely much" and another scale of taking test formulation again with 0="Never - under no circumstances" and 10= "Yes, definitely".

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom